CLINICAL TRIAL: NCT05904041
Title: Relationship Between E-health Literacy and Healthy Lifestyle Behaviors of University Students Studying Health Education in Turkey
Brief Title: E-health Literacy and Healthy Lifestyle Behaviors of University Students Studying Health Education in Turkey
Status: Completed | Type: Observational
Sponsor: KTO Karatay University (Other)
Responsible Party: Principal Investigator, Hasan Gerçek, Lecturer, KTO Karatay University
Other Study IDs: KaratatUH9
Record Dates: First submitted 2023-06-06; First posted 2023-06-15 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: E-health Literacy; Healthy Lifestyle Behaviors

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to examine the relationship between e-health literacy and healthy lifestyle behaviors of university students receiving health education in Turkey.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the study,
* being at least an associate degree student in the study area of health education

Exclusion Criteria:

* having any vision and hearing problems

Ages: 17 Years to 27 Years | Sex: All
Age Groups: Child, Adult
Study Population: University students
Sampling Method: Non-Probability Sample
Enrollment: 1454 (Actual)
Dates: Start 2023-06-06 (Actual); Primary Completion 2023-06-20 (Actual); Study Completion 2023-06-21 (Actual)

PRIMARY OUTCOMES:
E-health literacy | baseline
  The E-Health Literacy Scale will used to determine the participants' e-health literacy.The scale consists of 2 items related to internet use and 8 items measuring internet attitude. The scale items are organized as "1= strongly disagree, 2= disagree, 3= undecided, 4= agree, 5= strongly agree" with a 5-point Likert-type scaling method. The lowest score is 8 points and the highest score is 40 points. A high score obtained from the scale indicates a high level of e-health literacy.
Healthy lifestyle behavior | baseline
  Participants' healthy lifestyle behaviors were assessed with the Healthy Lifestyle. Behaviors Scale II The scale consists of 52 items and six factors. These are health responsibility, physical activity, nutrition, spiritual development, interpersonal relationships and stress management. The scale is scored on a scale of never=1, sometimes=2, often=3, regularly=4. A high score indicates relatively positive healthy living behaviors. The lowest score for the whole scale is 52 and the highest score is 208. The score of the whole scale gives the score of the healthy lifestyle behaviors. Higher scores indicate that the person practices the specified health behaviors at a high level

CONTACTS AND LOCATIONS:
Locations (1):
- KTO Karatay University, Konya, Karatay, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided